CLINICAL TRIAL: NCT02921035
Title: A Multicenter, Prospective, Non-interventional Study to Assess Adherence to Treatment for patIeNts With RMS Who Are Prescribed Subcutaneous (sc) Interferon Beta-1a (MAIN-MS)
Brief Title: Non-interventional Study to Assess Adherence to Treatment for Patients With RMS (MAIN-MS)
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Middle East FZ LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MS200136_0035
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Relapsing Multiple Sclerosis (RMS)
Keywords: Relapsing Multiple Sclerosis; Interferon beta-1a; Rebif®; Morisky Green Levine Medication Adherence Scale
MeSH Terms: interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relapsing Multiple Sclerosis (RMS) group: Subjects diagnosed with RMS who are prescribed Rebif (Interferon beta-1a)
  Interventions: Drug: Rebif (Interferon beta-1a)

INTERVENTIONS:
Drug: Rebif (Interferon beta-1a) — Rebif will be administered at a dose of 44 mcg, sc, tiw.

SUMMARY:
This is an open label, non randomized, uncontrolled, multicenter, single arm observational study. In this study, the enrolled subjects will be treated with Rebif human serum albumin (HSA)-free formulation (with or without RebiSmart) 44 microgram (mcg), subcutaneous (sc), thrice in a week (tiw) for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged more than or equal to (>=) 18 years and less than or equal to (<=) 60 years at the time of Rebif introduction
* Subjects diagnosed with RMS according to the revised McDonald criteria (2010)
* Treatment naïve or subjects on other DMDs who will switch to Rebif.
* Subjects will receive 1st Rebif 44 mcg dose after signing informed consent
* Subjects willing and able to provide signed informed consent.

Exclusion Criteria:

* Have any contraindications to treatment with IFN beta-1a sc according to European summary of product characteristics (EU SPC)/prescribed information
* Subjects participating in other clinical studies/trials
* Any female subject of childbearing potential who is not on contraceptives
* Subjects refusal to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects diagnosed with RMS and who are treatment naïve or on other disease modifying drugs (DMDs) will be enrolled into the study.
Sampling Method: Probability Sample
Enrollment: 594 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Percentage adherence of subjects on Rebif, using the Morisky Green Levine Medication Adherence Scale (MGLS) Score | Month 24
  MGLS is a four item self-reported questionnaire to assess medication adherence. It consists of four questions/items evaluating drug intake habits in subjects on chronic therapies with a scoring scheme of "Yes" = 1 (no adherence) and "No" = 0 (adherence). The items are summed to give an overall score, which ranges from 0 to 4 where high adherence=0, medium adherence=1-2 or low adherence=3-4.

SECONDARY OUTCOMES:
Percentage of subjects on Rebif who discontinued the treatment | up to 24 months
Time to treatment discontinuation | up to 24 months
Reason for treatment discontinuation | up to 24 months
  The reason for treatment discontinuation will includes: adverse event, lost to follow-up, lack of efficacy, protocol noncompliance, progressive disease, withdrew consent, death, frequency, unrealistic expectations, other
Percentage of relapse-free subjects | Month 24
Percentage of subjects with expanded disability status scale (EDSS) progression | Month 24
  EDSS is used for multiple sclerosis disability assessment. It is a 10 point scale, where 0 indicates normal motor skills, and 10 indicates patient's death. EDSS progression is defined as one point increase sustained for at least three months.
Number of subjects with suspected adverse drug reactions (ADRs) related to Rebif treatment and concomitant therapy over the 24 months of the study | Up to 24 months
Percentage of relapse-free subjects based on MGLS Score | Up to 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Merck Serono Middle East FZ-LLC, Study Director — an affiliate of Merck KGaA, Darmstadt, Germany
Locations (41):
- Algeria (6):
  - Research site, Algiers
  - Research site, Annaba
  - Research site, Blida
  - Research site, Oran
  - Research site, Sétif
  - Research site, Tizi Ouzou
- Argentina (3):
  - Research site, Mendoza
  - Research site, Rosario
  - Research site, San Miguel de Tucumán
- Research site, Manama, Bahrain
- Research site, Sofia, Bulgaria
- Egypt (4):
  - Research site, Al Mansurah
  - Research site, Alexandria
  - Research site 1, Cairo
  - Research site 2, Cairo
- Hungary (4):
  - Research site 1, Budapest
  - Research site 2, Budapest
  - Research site 3, Budapest
  - Research site, Esztergom
- Iran (2):
  - Research site, Isfahan
  - Research site, Tehran
- Research site, Kuwait City, Kuwait
- Lebanon (2):
  - Research site 1, Beirut
  - Research site 2, Beirut
- Morocco (6):
  - Research site, Casablanca
  - Research site, Fés
  - Research site, Marrakesh
  - Research site 1, Rabat
  - Research site 2, Rabat
  - Research site 3, Rabat
- Poland (6):
  - Research site, Gdansk
  - Research site, Katowice
  - Research site, Lodz
  - Research site, Lublin
  - Research site, Rybnik
  - Research site, Warsaw
- Saudi Arabia (4):
  - Research site, Dammam
  - Research site, Jeddah
  - Research site, Khober
  - Research site, Riyadh
- Research site 2, Seoul, South Korea

REFERENCES:
- [Derived] Al-Roughani R, Zakaria M, Cupler EJ, Taha K. Adherence to subcutaneous interferon beta-1a treatment among patients with relapsing multiple sclerosis: the MAIN-MS study. Front Neurol. 2023 Nov 28;14:1257455. doi: 10.3389/fneur.2023.1257455. eCollection 2023. PMID 38090266
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200136_0035
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html